CLINICAL TRIAL: NCT06997965
Title: An Open-label Single-arm Study to Assess the Efficacy of Mirikizumab in Patients With Inflammatory Strictures Due to Crohn's Disease
Brief Title: Open-label Single-arm Study to Assess the Efficacy of Mirikizumab in Patients With Inflammatory Strictures Due to CD
Acronym: MIRIAD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alimentiv Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELI-02022
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — mirikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mirikizumab (Other): Open-label mirikizumab 900mg IV Weeks 0,4, and 8 then mirikizumab 300mg SC Weeks 12, 16, 20, and 24.
  Interventions: Drug: Mirikizumab

INTERVENTIONS:
Drug: Mirikizumab — Mirikizumab is an IL-23 antagonist.
  Other Names: Omvoh

SUMMARY:
This is an open-label, single-arm, phase 4 study to assess the safety and efficacy of mirikizumab in approximately 60 participants with stricturing CD.

DETAILED DESCRIPTION:
This is an open-label, single-arm, phase 4 study to assess the safety and efficacy of mirikizumab in approximately 60 participants with stricturing CD. This study will enroll adults (≥18 years of age) with a diagnosis of ileal or ileocolonic CD based upon radiologic, clinical, endoscopic, and histologic evidence with tolerable obstructive stricture symptoms. Participants will be recruited from approximately 15 sites in 2 countries (United States and Canada).

This study consists of 3 study periods (screening period, open-label treatment period, and safety follow-up). After signing informed consent, potential study participants will be screened over a 5-week screening period, including MRE and ileocolonoscopy to confirm the presence of inflammatory strictures. Eligible participants will receive 900 mg mirikizumab IV Q4W to Week 12 and then 300 mg mirikizumab SC Q4W to Week 24.

During screening and Week 24 visits, participants will undergo MRE for blinded MRE disease activity assessment with the MaRIA score and assessment of stricture features. At the same time points, ileocolonoscopy with biopsy collection (2 from the ileum, 2 from the rectum, and 2 from each colonic segment [ascending, transverse, descending, and sigmoid]; 12 biopsies total) will be performed for blinded endoscopic and histopathologic disease activity assessments with the SES-CD and RHI, respectively.

Throughout the study, participants will undergo routine safety assessments at clinic visits, which will include physical examination, vital signs, clinical laboratory assessment, and recording of SAEs. At specified time points throughout the study, participants will complete a 7 day paper study diary consisting of patient reported items of the CDAI, UNRS, PGI-C, PGI-S, and the S-PRO. Blood samples will be collected at Weeks 12 and 24 for safety laboratory and CRP assessments. Stool samples will be collected at baseline and Week 24 for assessing FCP levels. The SIBDQ will be completed in-clinic at screening and Week 24.

Participants will undergo a Safety Follow-up Visit 4 weeks after the last dose of study treatment for safety assessments and recording of SAEs, severe liver injury (ALT or AST ≥ 3 × ULN), serious infections, and CD-related complications. The safety follow-up visit can be performed by telephone, unless the participant has any ongoing AEs that require follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Nonpregnant, nonlactating adults, ≥ 18 years of age.
2. Diagnosis of ileal or ileocolonic CD based on standard clinical, endoscopic, and histologic evidence; established at least 3 months prior to screening.
3. Presence of at least 1 inflammatory stricture in the terminal ileum* within reach of an endoscope (passable or nonpassable). Strictures should be noncritical, naïve or anastomotic stricture(s), caused by CD and confirmed centrally by MRE according to the following criteria:

   * Localized luminal narrowing (luminal diameter ≤ 50% relative to normal adjacent bowel); AND
   * Bowel wall thickening (≥ 25% relative to adjacent bowel; AND
   * Either prestenotic dilation (defined as a luminal diameter ≥ 3 cm) or nonpassable with adult colonoscope *Note: The terminal ileum is defined as the last 15 cm of ileum proximal to the ileocecal valve or ileocolonic anastomosis. Other small bowel strictures will be considered on a case-by-case basis following discussion with the sponsor. Two strictures within 3 cm are considered the same stricture, and a long segment with multiple areas of narrowing or multiple strictures, that have inflammation between them, is counted as 1 stricture.
4. Abdominal pain after eating and/or limitations in the amount/types of food eaten.
5. Presence of tolerable obstructive symptoms and not expected to require hospitalization, endoscopic balloon dilation, surgical resection, or additional therapy during the study period. Participants should have sufficient food intake, even with diet modification, defined as a stable weight over 4 weeks prior to initiation of study intervention.
6. Participants taking oral corticosteroids (eg, ≤ 20 mg/day prednisone or ≤ 9 mg/day budesonide) for ≥ 4 weeks prior to screening. Participants must be willing to undergo corticosteroid taper 8 weeks after initiation of study intervention as per standard of care.
7. Participants can be on stable background therapy for CD and must agree to maintain the background therapy during the study. Acceptable stable background therapies include:

   * Oral 5-ASA drugs or sulfasalazine ≤ 4.8 g per day, for ≥ 4 weeks prior to screening
   * AZA, 6-MP, or MTX for ≥ 4 weeks prior to Screening
   * Any rectal therapy for treatment of CD for ≥ 4 weeks prior to screening
   * Antidiarrheal drugs for ≥ 8 weeks prior to screening
   * Bile acid sequestrants for ≥ 4 weeks prior to screening
8. Contraceptive use by study participants should be in accordance with the mirikizumab product monograph and local guidelines.
9. Signed informed consent.

Exclusion Criteria:

1. History or current diagnosis of UC, indeterminate colitis, ischemic colitis, nonsteroidal anti inflammatory drug-induced colitis, idiopathic colitis (ie, colitis not consistent with CD), radiation colitis, microscopic colitis, colonic mucosal dysplasia, or untreated bile acid malabsorption.
2. CD-related complications:

   * Previous extensive small bowel resection, ileorectal anastomosis, or a proctocolectomy, with no more than 2 segments missing.
   * Short bowel syndrome.
   * Ileostomy (diverting or end), colostomy, small bowel stoma, or ileoanal pouch.
   * Inactive fistulae in or adjacent to an ileal stricture. Participants with perianal fistulae could be included provided there is no evidence of peri-anal abscess > 2 cm.
   * Suspected or diagnosed active intra-abdominal or perianal abscess that has not been appropriately treated.
   * Abscess located < 2 cm in relation to the stricture.
   * Toxic megacolon.
3. Any major surgery, in the investigator's opinion, performed within 8 weeks prior to screening or planned during the study (ie, any surgical procedure requiring general anesthesia).
4. Malignancies or history of malignancy within 5 years of the initial screening visit, except for adequately treated or completely excised nonmetastatic basal cell carcinoma, squamous cell carcinoma of the skin, or cervical carcinoma in situ.
5. Diagnosis of decompensated liver disease, including but not limited to autoimmune liver disease, viral hepatitis, Wilson disease, or suspected drug-induced liver injury.
6. Liver chemistry parameters that exceed the following thresholds:

   * ALT or AST > 2 × ULN
   * Alkaline phosphatase > 2.5 × ULN
   * Total bilirubin > 1.5 × ULN
7. Concomitant use of the following medications during the screening period or throughout the study:

   * Cyclosporine, tacrolimus, sirolimus, or mycophenolate mofetil within 8 weeks prior to screening.
   * Biologics (anti-tumor necrosis factor, anti-integrins, ustekinumab, or risankizumab) within 8 weeks prior to screening.
   * JAK inhibitor within 4 weeks prior to screening and throughout the study.
   * IL23p19 inhibitor within 4 weeks (or 5 half-lives, whichever is longer) prior to screening, or a history of nonresponse or intolerance to IL23p19 inhibitors.
8. Not up-to-date with current age-appropriate vaccinations in accordance with current immunization guidelines and the investigator's usual standard of care at screening.
9. Concurrent or previous participation in another clinical trial and received investigational therapy within 4 weeks or 5 half-lives (whichever is longer) prior to screening.
10. Any previous treatment with an antifibrotic therapy, including investigational antifibrotic therapies.
11. Systemic or opportunistic infections including:

    * HIV or hepatitis B or C infection. If a negative test result is available in the 12 months prior to Day 0, retesting is not required.
    * Known active or latent TB; if a negative test result is available in the 12 months prior to randomization, confirmatory testing (per standard of care) is not required before Day 0.
    * Positive stool test for Clostridioides difficile infection (as demonstrated by positive toxin).
    * Active CMV infection, as per investigator judgement
    * Other systemic or opportunistic infection, any other clinically significant extraintestinal infection, infection that is not responding to standard treatment, or recurring infection within 6 months of Day 1.
12. Known or suspected allergy, anaphylaxis, hypersensitivity or intolerance to mirikizumab or its' excipients.
13. Contraindication to MRE examination or suspected allergy to MRE contrast agent or antispasmodic.
14. Prior enrolment in the current study and had received study treatment.
15. Any acute or chronic medical condition, psychiatric disorder, or laboratory abnormality that may increase the risk associated with study participation or study intervention administration, or may interfere with the interpretation of study results, as determined by the investigator.
16. Unwillingness to withhold protocol-prohibited medications during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of mirikizumab in inducing a radiologic response in participants with inflammatory stricturing CD | At week 24
  Achievement of radiologic response (defined by a ≥ 50% improvement in stricture length and no worsening of prestenotic small bowel diameter OR a ≥ 50% improvement in prestenotic small bowel diameter and no worsening of stricture length)

SECONDARY OUTCOMES:
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 4
  Change from baseline in S PRO score
To evaluate the efficacy of mirikizumab in health-related quality of life in participants with inflammatory stricturing CD | At week 4
  Change from baseline in S PRO score
To evaluate the efficacy of mirikizumab in radiologic disease activity in participants with inflammatory stricturing CD | At week 4
  Change from baseline in S PRO score
To evaluate the efficacy of mirikizumab in endoscopic disease activity in participants with inflammatory stricturing CD | At week 4
  Change from baseline in S PRO score
To evaluate the efficacy of mirikizumab in histologic disease activity in participants with inflammatory stricturing CD | At week 4
  Change from baseline in S PRO score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 8
  Change from baseline in S PRO score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 12
  Change in baseline in S PRO score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 16
  Change from baseline in S PRO score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 20
  Change from baseline in S PRO score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 24
  Change from baseline in S PRO score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 12
  Change from baseline in CDAI score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 24
  Change from baseline in CDAI score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 12
  Change from baseline in PRO2 Score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 24
  Change from baseline in PRO2 score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 12
  Change from baseline in HBI score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 24
  Change from baseline in HBI score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 24
  Achievement of endoscopic response (defined by ≥ 50% reduction from baseline in SES-CD score) AND radiographic improvement (defined by a ≥ 25% improvement from baseline in stricture MaRIA score)
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 24
  Achievement of endoscopic response (defined by ≥ 50% reduction from baseline in SES-CD score)
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 24
  Change from baseline in SIBDQ score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 12
  Change from baseline in UNRS score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 24
  Change from baseline in UNRS score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 24
  Change from baseline in RHI score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 24
  Achievement of histological response (defined by a ≥ 50% reduction from baseline in RHI score)
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 12
  Achievement of CRP response (defined by ≥ 50% reduction from baseline in CRP levels)
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 24
  Achievement of CRP response (defined by ≥ 50% reduction from baseline in CRP levels)
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 12
  Change from baseline in CRP level
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 24
  Change from baseline in CRP level
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 24
  Achievement of FCP response (defined by ≥ 50% reduction from baseline in FCP level)
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 24
  Change from baseline in FCP level
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 4
  Change from baseline in PGI-S score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 8
  Change from baseline in PGI-S score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 12
  Change from baseline in PGI-S score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 16
  Change from baseline in PGI-S score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 20
  Change from baseline in PGI-S score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 24
  Change from baseline in PGI-S score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 4
  PGI-S score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 8
  PGI-S score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 12
  PGI-S score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 16
  PGI-S score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 20
  PGI-S score
To evaluate the efficacy of mirikizumab in improving symptoms in participants with inflammatory stricturing CD | At week 24
  PGI-S score
To evaluate the safety of mirikizumab in participants with stricturing CD | Through end of safety follow-up
  Occurrence of SAEs, severe liver injury (ALT or AST ≥ 3 × ULN), and serious infections
To evaluate the safety of mirikizumab in participants with stricturing CD | Through end of safety follow-up defined as a composite of (1) CD-related surgery, (2) CD-related hospitalization, (3) CD-medication-related complication, and (4) rescue therapy for a documented CD-related flare
  CD-related complications